CLINICAL TRIAL: NCT06984861
Title: Major Radiation Dose De-Escalation Concurrent With Chemotherapy for Advanced Stage Human Papilloma Virus Associated Oropharyngeal Carcinoma
Brief Title: A Study of Reduced Radiation Therapy With Chemotherapy in People With HPV-Positive Throat Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-040
Record Dates: First submitted 2025-05-14; First posted 2025-05-22 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Oropharyngeal Carcinoma
Keywords: Human Papilloma Virus Associated; Chemoradiation; T3-4/N0-2c or any N3; 25-040
MeSH Terms: conditions — Oropharyngeal Neoplasms | interventions — Chemoradiotherapy; Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: This non-randomized phase II study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Radiation Therapy With Chemotherapy in People With HPV-Positive Throat Cancer (Experimental): Subjects will first undergo 6 weeks of standard induction chemotherapy and if downstaged to T1-2 and <N3 and also have no evidence of hypoxia will undergo a major de-escalated radiation therapy to 30Gy concurrent with standard chemotherapy. Hypoxia status is determined by the absence of hypoxia uptake on Fluorine-18-Labeled Fluoro-Misonidazole (18F-FMISO) PET/CT imaging (8-10 treatment days after start of chemoradiation), which has an FDA approved IND for use in humans . If the 18F-FMISO PET is negative for hypoxia, the patient will receive 30Gy concurrent with 2 cycles of chemotherapy. If the 18F-FMISO PET is positive for hypoxia, the patient will receive standard of care 70Gy concurrent with 3 cycles of chemotherapy.
  Interventions: Diagnostic Test: 18F-FMISO PET/CT Scan; Combination Product: Chemoradiation; Other: Questionnaires

INTERVENTIONS:
Diagnostic Test: 18F-FMISO PET/CT Scan — The 18F-FMISO PET/CT Scan Protocol consists first of an IV bolus injection of approximately 5-10 mCi of the radiotracer. Subjects will undergo 18F-FMISO scan (only 1 injection) occurs at 8-10 treatment days* into chemoradiation. Each patient will have a baseline staging FDG PET scan which is used to localize the tumor at the primary site and all suspicious cervical neck nodes (> 1 cm in short axis diameter with focal abnormal increased FDG avidity). These lesions are then assessed on the respective 18F-FMISO PET/CT.
Combination Product: Chemoradiation — Patients will start with induction chemotherapy of carboplatin, paclitaxel and cetuximab for 6 weeks and when downstaged to T1-2 and < N3, the patient is eligible to receive concurrent chemoradiation per protocol.A total radiation therapy of 30Gy will be delivered to the oropharynx and neck at 2Gy per fraction per day over 15 days for patients who exhibited no evidence of hypoxia on the intra-treatment 18F-FMISO PET/CT. Concurrent chemotherapy (2 cycles) will be given. After completion of chemotherapy and radiation therapy, a 4 month (+/- 4 weeks)
Other: Questionnaires — EQ-5D-5L, MDADI-HN, COST-FACIT

SUMMARY:
The researchers are doing this study is to find out if lower doses (given in fewer treatments over a shorter period of time) of radiation therapy in combination with standard-of-care chemotherapy is an effective treatment for people with Human Papilloma Virus (HPV)-positive throat cancer and works as well as the standard doses of radiation therapy in combination with standard-of-care chemotherapy. The chemotherapy drugs used in combination with radiation therapy in this study include cisplatin, carboplatin, and 5-fluorouracil (5-FU).

ELIGIBILITY:
Inclusion Criteria:

* Pathologically (histologically or cytologically) proven diagnosis of HPV associated squamous cell carcinoma of the oropharynx (tonsil, base of tongue, or oropharyngeal walls) from biopsy, surgical resection or excisional biopsy regardless of margin status.

  1. Squamous cell carcinoma of the neck of unknown primary is allowed with excision biopsy of a lymph node (or core biopsy) or consent from the PI or co-PI. Patient must have excisional biopsy or core biopsy done in order to be on protocol.

     Note: Evidence of HPV associated oropharyngeal cancer from either the primary tumor site or from a lymph node. A patient is HPV positive when he or she tests positive having tested positive for both p16 expression (70% nuclear and cytoplasm expression; Ventana Medical Systems) and mRNA HPV in situ hybridization.
* Subjects must have clinically or radiographically evident measurable gross disease at either the primary tumor site or nodal stations.
* Oropharyngeal Carcinoma (AJCC, 7th ed.) without evidence of distant metastasis based on FDG PET/CT.
* CT or MRI of the neck with and without contrast Note: A CT scan of neck and/or a PET/CT performed for the purposes of radiation planning may serve as planning tools.
* ECOG Performance Status of 0-2 or KPS ≥ 70
* Age ≥ 18
* Adequate hematologic function within 30 days prior to registration, defined as follows:

  1. White Blood Count (WBC) ≥ 2 K/mcL
  2. Absolute neutrophil count (ANC) ≥ 1,000 cells/mm^3
  3. Platelets ≥ 100,000 cells/mm^3
  4. Hemoglobin ≥ 8.0 g/dl

Note: The use of transfusion or other intervention to achieve Hgb ≥ 8.0 g/dl is acceptable

* Adequate renal function within 30 days prior to registration, defined as follows:

  a. Serum creatinine ≤ 1.5 mg/dl or creatinine clearance (CC) ≥ 50 ml/min determined by 24-hour collection or estimated by Cockcroft-Gault formula CCr male = [(140 - age) x (wt in kg)] [(Serum Cr mg/dl) x (72)] CCr female = 0.85 x (CrCl male) Note: Patients who cannot tolerate cisplatin or carboplatin/5FU based on clinical judgment will receive carboplatin and paclitaxel
* Adequate hepatic function within 30 days prior to registration, defined as follows:

  1. Bilirubin ≤ 2 mg/dl
  2. AST or ALT ≤ 3 x the upper limit of normal Note: Patients who cannot tolerate cisplatin or carboplatin/5FU based on clinical judgment will receive carboplatin and paclitaxel. Negative serum pregnancy test within 14 days prior to registration for women of childbearing potential
* The subject must provide study-specific informed consent prior to study entry Subject able to undergo MRI scans except for major medical contraindications like presence of a pacemaker or approved by the PI or the CO-PI that the subject does not need to undergo MRI scans

Exclusion Criteria:

* Subjects with prior head and neck radiation therapy
* Subjects with simultaneous primary cancers outside of the oropharynx if determined by the PI/Co-PI the patient can proceed with protocol activities.

Note: Exceptions can be made for patients with simultaneous primaries outside the oropharynx if determined by the PI/Co-PI the patient can proceed with protocol activities.

* Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for 3 years or if cure rate from treatment at 5 years to be 90% or greater
* Prior systemic chemotherapy for the study cancer; note that prior chemotherapy for a different cancer is allowable
* Severe, active co-morbidity defined as follows (exceptions can be made if approved by the PI and/or co-PI)

  1. Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months
  2. Transmural myocardial infarction within the last 6 months
  3. Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
  4. Chronic Obstructive Pulmonary Disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy within 30 days of registration
  5. Hepatic Insufficiency resulting in clinical jaundice and/or coagulation defects

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2025-05-13 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Locoregional control | 2 years
  Researchers will test the null hypothesis H0: P=78% vs the alternative hypothesis H1:P=91%, where P represents the 2-year locoregional control (LRC). We will use the Kaplan-Meier method to estimate the LRC rate at 2 years and construct a 0.975 1-sided confidence interval in order to achieve a test size alpha = 0.05 (this is based on a finite-sample correction using 100,000 simulations).

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Lee, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk- Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org